CLINICAL TRIAL: NCT04829617
Title: A Novel Behavioral Intervention to Promote Adherence in Heart Failure
Brief Title: Promoting Well-being and Health in Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Christopher Celano, Psychiatrist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021P000882
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Heart Failure NYHA Class I; Heart Failure NYHA Class II; Heart Failure NYHA Class III
Keywords: Positive Psychology; Physical Activity; Low-Sodium Diet; Medication Adherence; Motivational Interviewing
MeSH Terms: conditions — Heart Failure; Motor Activity; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded, controlled trial
Who Masked: Outcomes Assessor
Masking Description: Participants and treating study staff will be aware of the participant's treatment condition. However, follow-up assessments will be performed by a study staff member that is masked to the participant's treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PP-MI Intervention (Experimental): Participants will receive a 12-week, Positive Psychology-Motivational Interviewing (PP-MI) intervention. Each week, participants will complete a PP activity and work towards one or more health behavior goals, then complete a phone session with a study trainer. Each weekly session will include PP and goal setting portions. In the PP portion, a study trainer will (a) review the week's PP exercise, (b) discuss the rationale of the next week's PP exercise through a guided review of the PP-MI manual, and (c) assign the next week's PP exercise. Additionally for the goal-setting portion, the trainer will (a) review their goals and health behaviors from the prior week, (b) discuss techniques for improving health behavior adherence (e.g., monitoring physical activity, reading nutrition labels), and (c) set goals for the next week. Finally, participants will receive supplemental text messages throughout the 12 weeks of the intervention and during the initial follow-up period (Week 13-24).
  Interventions: Behavioral: PP-MI Intervention
- MI-alone Intervention (Active Comparator): This condition will mirror the MI component of the PP-MI intervention. During the first three sessions, participants will learn about the causes and types of HF, risk factors for cardiovascular disease, and methods for monitoring risk factors and symptoms. Then participants will complete nine sessions related to physical activity, a low sodium diet, and medication adherence. Weekly tasks (e.g., brainstorming barriers) will be assigned, completed between calls, and reviewed at the following call. Finally, participants will receive supplemental text messages throughout the 12 weeks of the intervention and during the initial follow-up period (Week 13-24).
  Interventions: Behavioral: MI-alone Intervention

INTERVENTIONS:
Behavioral: PP-MI Intervention — The 12-week PP-MI intervention focuses on enhancing well-being (through PP) and promoting adherence to physical activity, diet, and medications (through MI). Each week, participants will complete a PP activity and work towards one or more health behavior goals, then complete a phone session with a study trainer. The PP portion of the program will focus on the cultivation of well-being through the performance of easy-to complete activities (e.g., using a strength in a new way) and review of the positive feelings they generate. The MI portion of the program will focus on assisting participants to monitor health behavior adherence, resolve ambivalence to behavior change, set realistic health behavior goals, problem-solve barriers, and identify resources to complete behavior change. Finally, participants will receive twice weekly text messages (for 24 weeks) to encourage completion of PP activities and engagement in health behaviors.
  Arms: PP-MI Intervention
Behavioral: MI-alone Intervention — The time- and attention-matched MI-alone intervention focuses on providing education about heart failure (HF) and promoting adherence to physical activity, diet, and medications. Each week, participants will independently complete an activity related to HF education or adherence to a health behavior, then complete a phone session with a study trainer. HF educational topics will include the causes and types of HF, risk factors for cardiovascular disease, methods for monitoring risk factors and symptoms, and the importance of adherence to physical activity, diet, and medications. For each health behavior, study trainers will assist participants to monitor adherence, identify realistic behavior goals, problem-solve barriers, and identify resources to complete behavior change. Finally, participants will receive twice weekly text messages (for 24 weeks) that provide education and encourage engagement in health behaviors.
  Arms: MI-alone Intervention

SUMMARY:
The focus of this study is to test the efficacy of a 12-week, phone-delivered Positive Psychology-Motivational Interviewing (PP-MI) intervention, with additional twice weekly PP and health behavior text messages for a total of 24 weeks (with interactive, algorithm-driven, goal-focused text messages in the final 12 weeks), compared to an attention-matched MI-based educational condition, in a randomized trial (NIH Stage II) of 280 patients with New York Heart Association class I-III Heart Failure (HF).

DETAILED DESCRIPTION:
The investigators are proposing a study that will focus on testing the efficacy of a Positive Psychology-Motivational Interviewing (PP-MI) intervention, with additional twice weekly PP and health behavior text messages for a total of 24 weeks (with interactive, algorithm-driven, goal-focused text messages in the final 12 weeks) in patients with New York Heart Association class I-III HF. The investigators will enroll 280 HF patients, who will take part in a 12-week (with 24 weeks of supplemental text messages) health behavior intervention.

In this project, the investigators hope to do the following:

1. Examine the efficacy of a 12-week, phone-delivered PP-MI intervention for individuals with heart failure (HF) on health behavior adherence at 12 weeks (primary time point), 24 weeks, and 48 weeks.
2. Assess the intervention's impact on psychological outcomes, health-related quality of life (HRQoL), HF-specific quality of life, HF symptoms, and function.
3. Explore the intervention's impact on markers of cardiovascular health (e.g., blood pressure), as well as major adverse cardiac events, HF hospitalizations, and mortality.

Participants will undergo two visits (in-person or virtual) during which they will meet with study staff. During the first visit, participants will provide informed consent, answer questionnaires related to psychological and physical health and functioning, have their blood pressure and weight measured, and be asked to monitor their physical activity (using an accelerometer) for one week and medication adherence (using an electronic pill bottle) for two weeks. Participants will be given a urine collection container and asked to provide a urine sample within 4 hours of their first void and before eating breakfast on the day of Visit 2. At the second visit, the urine sample will be collected, and upon confirmation of adequate physical activity and medication adherence data, participants will be randomized to receive the PP-MI intervention or the MI-alone intervention.

Following randomization, all participants will be provided a treatment manual corresponding with their treatment condition, a Fitbit activity tracker, and other treatment materials. The appropriate intervention will be introduced, and the first exercise will be assigned.

Following the second visit, participants in both treatment conditions will complete twelve weekly phone sessions with a study trainer. The phone sessions primarily will include a review of the prior week's session content and a discussion of the rationale and assignment of the next week's exercise/assignment.

Participants in both treatment conditions will receive twice weekly text messages throughout the intervention (Weeks 1-12) and initial follow-up period (Weeks 13-24). During the intervention, these messages will provide information about the PP activity (PP-MI group) and health behavior goal (both groups) discussed that week. During Weeks 13-24, participants in the PP-MI condition will engage with twice weekly, automated, interactive text messages related to PP and health behavior goals. Individuals in the MI-alone group will receive identical messages related to setting health behavior goals as the PP-MI participants and will additionally receive a fixed test message providing education about health behavior adherence.

At Weeks 12, 24, and 48, participants will complete follow-up visits. One week prior to these visits, participants will be mailed an accelerometer and will wear it until their study visit. They will also be sent a container for urine collection, which they will bring to their follow-up visit. During these study visits, participants will be asked to answer questionnaires related to psychological and physical health and functioning, have their blood pressure, weight, and waist circumference measured, will perform a 6 minute walk test, and be asked about cardiovascular outcomes, including hospitalizations, cardiovascular procedures, and cardiac-specific hospitalizations.

Finally, participants will complete phone sessions every 6 months until study end to inquire about hospitalizations and adverse cardiac events.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with NYHA class I, II, or III HF.
* Suboptimal adherence to health behaviors. This will be defined as a total score of ≤15 on three Medical Outcomes Study Specific Adherence Scale (MOS) items regarding diet/exercise/medications.

Exclusion Criteria:

* Cognitive deficits impeding a participant's ability to provide informed consent or participate, assessed via a 6-item cognitive test.
* Medical conditions likely to lead to death within 6 months.
* Inability to participate in physical activity due to another medical condition (e.g., arthritis).
* Inability to read, write, or speak in English.
* Current participation in another intervention or program that has been designed to promote well-being or health behavior adherence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Health behavior adherence | Baseline, 12 Weeks, 24 Weeks, 48 Weeks
  Composite score of overall activity (measured by accelerometer in steps/day), sodium excretion (urine sodium in mEq/day), and medication adherence (Medication Event Monitoring System [MEMS] electronic pill bottle). This composite score will be created by calculating z scores for each individual outcome measure and then averaging them for each participant at each time point.

SECONDARY OUTCOMES:
Physical activity (in steps/day) | Measured for 7 days at baseline, 12 weeks, 24 weeks, and 48 weeks
  Physical activity (steps) will be measured via an accelerometer. We will use established accelerometer protocols to measure the mean number of steps taken per day at each time point.
Objective medication adherence (Medication Event Monitoring System [MEMS] pill bottles) | Measured for 14 days at baseline, 12 weeks, 24 weeks, and 48 weeks
  Medication adherence will be measured using MEMS electronic pill bottles. Participants will receive a MEMS pill bottle at the initial study visit and will be asked to put one cardiac medication (loop diuretic, ACE inhibitor, beta blocker, or aspirin, in that order) in the bottle and then use it throughout the study period (48 weeks). Adherence will be measured by the percentage of appropriate bottle openings over a 2-week period at baseline and the follow-up time points.
Sodium Excretion (mEq/day) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Objective sodium intake will be assessed through the measurement of urinary sodium excretion. Participants will provide a sample of their second voiding of the day, and from this sample, urine sodium and urine creatinine will be measured.
Positive Affect (Positive and Negative Affect Schedule [PANAS] positive affect items) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Positive affect will be measured using the 10 positive affect items from the PANAS, a well-validated scale used in numerous other behavioral intervention trials.
Physical Function (PROMIS 20-item Physical Function Short Form [PF-20]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  The PROMIS 20-item short form (PF-20) will be used to assess physical function.

OTHER OUTCOMES:
Moderate to Vigorous Physical Activity (MVPA) | Measured for 7 days at baseline, 12 weeks, 24 weeks, and 48 weeks
  MVPA (reported in mean minutes of MVPA/day) will be measured via an accelerometer and recorded in mean minutes/day.
Sedentary Time (mean minutes/day) | Measured for 7 days at baseline, 12 weeks, 24 weeks, and 48 weeks
  Sedentary time (mean minutes/day) will be measured via Actigraph accelerometer.
Self-reported sodium intake (Scored Sodium Questionnaire [SSQ]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  The Scored Sodium Questionnaire (SSQ) measures the frequency with which individuals have consumed sodium-containing foods in the past month.
Self-report medication adherence (tool from the NHLBI Heart and Soul Study) | Measured for 14 days at baseline, 12 weeks, 24 weeks, and 48 weeks
  Medication adherence will be measured with the self-report medication adherence tool from the NHLBI Heart and Soul Study.
Optimism (Life Orientation Test - Revised [LOT-R]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Optimism will be measured using the LOT-R, a frequently used 6-item instrument that assesses dispositional optimism.
Self-efficacy (General Self-Efficacy Scale [GSE]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Self-efficacy will be measured using the General Self Efficacy scale (GSE), a validated measure of self-efficacy, given its links to improved adherence.
Depressive symptoms (Hospital Anxiety and Depression Scale - depression subscale [HADS-D]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Depressive symptoms will be measured using the 7-item depression subscale of the HADS.
Anxiety (Hospital Anxiety and Depression Scale - anxiety subscale [HADS-A]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Anxiety will be measured using the 7-item anxiety subscale of the HADS.
Locus of control (Form C of the Multidimensional Health Locus of Control scale [MHLC Form C]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Locus of control will be measured using the 18-item MHLOC.
Health-related quality of life (Medical Outcomes Study Short Form-12 [SF-12]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  The SF-12 will be used to assess health-related quality of life. The SF-12 produces both mental and physical component scores, both of which will be assessed this trial.
HF-related quality of life (Kansas City Cardiomyopathy Questionnaire [KCCQ] quality of life score) | Baseline, 12 weeks, 24 weeks, 48 weeks
  HF-related quality of life will be assessed using the quality of life score from the KCCQ.
HF symptoms (Kansas City Cardiomyopathy Questionnaire [KCCQ] total symptom score) | Baseline, 12 weeks, 24 weeks, 48 weeks
  HF symptoms will be measured using the KCCQ total symptom score.
Systolic and diastolic blood pressure | Baseline, 12 weeks, 24 weeks, 48 weeks
  Blood pressure (diastolic and systolic) will be measured by trained nurses using a standardized protocol.
Body mass index | Baseline, 12 weeks, 24 weeks, 48 weeks
  Height and weight (for calculation of body mass index) will be measured by trained nurses.
Waist circumference | Baseline, 12 weeks, 24 weeks, 48 weeks
  Waist circumference will be measured by trained nurses and/or dieticians.
LDL and HDL cholesterol | Baseline, 12 weeks, 24 weeks, 48 weeks
  Fasting lipids (including LDL and HDL cholesterol) will be measured via blood samples.
Triglycerides | Baseline, 12 weeks, 24 weeks, 48 weeks
  Fasting lipids (including triglycerides) will be measured via blood samples.
Fasting blood glucose | Baseline, 12 weeks, 24 weeks, 48 weeks
  Fasting blood glucose levels will be measured via a blood sample.
6-minute walk test (in meters traveled) | Baseline, 12 weeks, 24 weeks, 48 weeks
  A 6-minute walk test will be measured and monitored by trained nurses and/or dieticians to measure functional capacity.
Major Adverse Cardiac Events (MACE) | Throughout study period (estimated mean duration 28 months)
  MACE will be defined as mortality or hospitalization for HF or an acute coronary event (percutaneous coronary intervention or acute coronary syndrome). Data regarding hospitalizations and mortality will be obtained using a three-pronged approach consisting of systematic queries of participants, electronic health record review, and review of records from the National Death Index.
All-cause Hospitalizations | Throughout study period (estimated mean duration 28 months)
  We will record all-cause hospitalizations for all participants from enrollment to the end of the study data collection period, using systematic queries of participants and review of electronic health records from all Mass General Brigham-affiliated hospitals.
Heart Failure Hospitalizations | Throughout study period (estimated mean duration 28 months)
  We will record HF hospitalizations for all participants from enrollment to the end of the study data collection period, using systematic queries of participants and review of electronic health records from all Mass General Brigham-affiliated hospitals.
Mortality | Throughout study period (estimated mean duration 28 months)
  We will record vital status for participants from enrollment to the end of study data collection. Data regarding mortality will be obtained using electronic health record review and review of records from the National Death Index.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Celano, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
To promote sharing of study data with other researchers, we also will create a deidentified study dataset. We will include both item-level and summary scores for each scale and will include data from the baseline, 12-week, 24-week, and 48-week time points.
Supporting Information: Study Protocol, SAP
Time Frame: This information will be shared prior to the end of the study funding period.
Access Criteria: Investigators who are interested in obtaining access to this information will be asked to submit a request to the principal investigator outlining the proposed use of the data and would need to agree to certain conditions (e.g., not attempting to identify individual participants, destroying data once the use of the data is complete) prior to obtaining access.